CLINICAL TRIAL: NCT06843356
Title: Trial of Rescue Endovascular Treatment for Progressive Acute Mild Ischemic Stroke With Basilar Artery Occlusion With Extended Time Window
Acronym: RESCUE-BAO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Wannan Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RESCUE-BAO
Record Dates: First submitted 2025-02-20; First posted 2025-02-24 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Acute Mild Ischemic Stroke; Basilar Artery Occlusion; Rescue Endovascular Treatment; Extended Time Window

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Endovascular Therapy Group (Experimental): Researchers can choose to deal with the stenosis or occlusion of blood vessels according to their own judgment, including stent thrombectomy, thrombus aspiration, balloon angioplasty, stent replacement, intra-arterial thrombolysis or various combinations of these methods.
  Interventions: Procedure: Endovascular Treatment
- Best Medical Management Group (No Intervention): Participants receive best medical management only. Best Medical Treatment and maximum supportive care according to local guidelines, not including mechanical thrombectomy, no intra-arterial treatment.

INTERVENTIONS:
Procedure: Endovascular Treatment — Neurointerventionist determine whether to proceed with interventional therapy after assessing the location and degree of occlusion, the tortuosity of the access vessel, and the presence of stenosis or occlusion in the proximal artery. In cases where there is no proximal stenosis or occlusion, mechanical thrombectomy is performed, and the specific thrombectomy strategy is tailored by the researcher based on the patient's condition. For lesions associated with proximal vascular stenosis or occlusion, it is necessary to navigate the catheter through the proximal stenosis or occlusion to access the intracranial occlusion. Researchers have the discretion to treat the stenotic or occluded vessels, which may include options such as no treatment, stent thrombectomy, thrombus aspiration, balloon angioplasty, stent replacement, intra-arterial thrombolysis or various combinations of these methods.
  Arms: Endovascular Therapy Group

SUMMARY:
A prospective, multicenter, open-label, blinded-endpoint, randomized controlled trial to evaluate whether best medical management (BMM) combined with endovascular therapy (EVT) improves neurological outcomes compared to BMM alone in patients with progressive acute mild ischemic stroke due to basilar artery occlusion within an extended time window.

DETAILED DESCRIPTION:
This trial aims to evaluate whether best medical management (BMM) combined with endovascular therapy (EVT) improves neurological outcomes compared to BMM alone in patients with progressive acute mild ischemic stroke due to basilar artery occlusion within an extended time window. The study used a stratified block randomization method, with stratification by center. A central randomization system was used to assign subjects to the experimental group and the control group in a 2:1 ratio for each center.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Symptoms and signs consistent with basilar artery ischemia.
3. Basilar artery or vertebral artery occlusion confirmed by computed tomography angiography (CTA), magnetic resonance angiography (MRA), or digital subtraction angiography (DSA); if vertebral artery occlusion is present, it should completely block blood flow along the basilar artery.
4. First-time onset meeting the criteria for mild ischemic stroke diagnosis: NIHSS score <6.
5. Symptom progression within 7 days of the first onset.
6. Symptom progression: NIHSS score increase ≥4 points or consciousness level increase ≥2 points from the initial NIHSS score.
7. Time from symptom onset to randomization >24 hours.
8. Symptom progression to randomization time ≤24 hours.
9. NIHSS score ≥10 before randomization.
10. pc-ASPECTS before randomization ≥ 6
11. The patient or their family members are willing to comply with the protocol requirements and data collection procedures, understand, and sign the informed consent form.

Exclusion Criteria:

1. Symptom progression due to intracranial hemorrhage, brain edema, or other clear causes (including but not limited to infarct hemorrhagic transformation, new infarction in non-occluded vascular regions, severe infection, high fever, heart or kidney dysfunction, hypovolemia, or severe electrolyte disturbances).
2. mRS >2.
3. Factors in the target vessel that are expected to prevent completion of endovascular treatment.
4. Multiple vessel occlusions.
5. Prior imaging confirmed or investigator-assessed chronic basilar artery occlusion.
6. Presence of untreated intracranial aneurysms, intracranial tumors (except small meningiomas), or intracranial vascular malformations.
7. Intracranial hemorrhage within the past 6 months, including parenchymal brain hemorrhage, intraventricular hemorrhage, or subarachnoid hemorrhage.
8. Gastrointestinal or urinary tract bleeding, acute myocardial infarction, cranial trauma, or major surgery within the past month.
9. Presence of active bleeding, coagulation disorders, or uncorrectable bleeding tendencies.
10. Platelet count <40×10^9/L, or INR >2 during anticoagulation therapy (irreversible).
11. Severe heart, liver, or kidney dysfunction or other severe systemic late-stage diseases.
12. Known allergy to iodine contrast agents or other treatment-related drugs.
13. Medically uncontrolled refractory hypertension (defined as persistent systolic blood pressure >185 mmHg or diastolic blood pressure >110 mmHg) (Note: Participants can be included if their blood pressure is controllable with medication and maintained at an acceptable level).
14. Uncontrollable blood glucose <2.8 mmol/L or >22.2 mmol/L.
15. Pregnancy or breastfeeding.
16. Life expectancy <6 months.
17. Participation in other clinical studies that may affect outcome assessment.
18. Investigator's judgment that the patient is unsuitable for participation in this study or may face significant risks (e.g., due to mental illness, cognitive, or emotional disorders preventing understanding and/or compliance with study procedures and/or follow-up).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with a modified Rankin Scale (mRS) score of 0-3 at 90 (±7) days after randomization. | 90 (±7)days after procedure
  The modified Rankin Score is an ordinal hierarchical scale ranging from 0 to 6, with higher scores indicating more severe disability.

SECONDARY OUTCOMES:
Shift analysis of the improvement trend in modified Rankin Scale (mRS) scores at 90 (±7) days after randomization. | 90 (±7) days after procedure
  Shift analysis is a statistical method used to evaluate the overall distribution change in modified Rankin Scale (mRS) scores, assessing whether an intervention leads to a general shift toward better outcomes across all score categories.
Proportion of patients with a modified Rankin Scale (mRS) score of 0-2 at 90 (±7) days after randomization. | 90 (±7) days after procedure
  The modified Rankin Score is an ordinal hierarchical scale ranging from 0 to 6, with higher scores indicating more severe disability.
Change in NIHSS score from baseline at 24 hours postoperatively. | 24 hours after procedure
  The NIHSS (National Institutes of Health Stroke Scale) is a tool used to assess the severity of stroke symptoms by evaluating various neurological functions, such as consciousness, vision, movement, and speech. The score helps in gauging the degree of impairment caused by a stroke.
EQ-5D-5L scale at 90 (±7) days after randomization. | 90 (±7) days after procedure
  The EQ-5D-5L scale is a standardized tool used to measure a person's health-related quality of life. It includes five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, each with five levels to indicate the severity of problems in those areas.
Change in NIHSS score from baseline at discharge or 5-7 days postoperatively. | Discharge or 5 -7 days after procedure.
  The NIHSS (National Institutes of Health Stroke Scale) is a tool used to assess the severity of stroke symptoms by evaluating various neurological functions, such as consciousness, vision, movement, and speech. The score helps in gauging the degree of impairment caused by a stroke.
Successful reperfusion postoperatively. | At the end of the operation
  The eTICI (extended Thrombolysis in Cerebral Infarction) score is a standard used to evaluate the degree of reperfusion in acute ischemic stroke patients following endovascular therapy (EVT). It is a further refinement of the mTICI (modified TICI) score.

OTHER OUTCOMES:
Incidence of symptomatic intracerebral haemorrhage (sICH) within 24 (±6) hours after randomization (Heidelberg bleeding classification). | Within 24 (±6) hours after procedure
  Intracranial hemorrhage (ICH) was assessed with the Heidelberg Bleeding Classification within 24 (±6) hours of endovascular treatment. Intracranial hemorrhage was classified as hemorrhagic infarction or parenchymal hematoma. The sICH was defined as ICH associated with a worsening of 4 or more points on the NIHSS or resulting in death, and cerebral herniation, which were not present at baseline.
Incidence of any intracerebral haemorrhage within 24 (±6) hours after randomization (Heidelberg bleeding classification). | within 24 (±6) hours after procedure
  Intracranial hemorrhage (ICH) was assessed with the Heidelberg Bleeding Classification within 24 (±6) hours of endovascular treatment. Intracranial hemorrhage was classified as hemorrhagic infarction or parenchymal hematoma.
All-cause mortality at 90 (±7) days after randomization. | 90 (±7) days after procedure
  All-cause mortality refers to the rate of death from any cause within a specific time period, without considering the underlying cause of death.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui, China